CLINICAL TRIAL: NCT00730912
Title: Protocol for Post-approval Commitment Study of Loratadine for PPK Analysis in Japanese Pediatric and Adults Patients
Brief Title: Post Approval Pharmacokinetic Study of Loratadine in Japanese Pediatric and Adult Patients (Study P05539)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: P05539
Record Dates: First submitted 2008-08-06; First posted 2008-08-08 (Estimated); Results first posted 2010-07-05 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-03

CONDITIONS: Perennial Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic, Perennial | interventions — Loratadine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Pediatrics 3 to 6 years (Experimental): Pediatrics 3 to 6 years
  Interventions: Drug: loratadine
- Pediatrics 7 to 15 years (Experimental): Pediatrics 7 to 15 years
  Interventions: Drug: loratadine
- Adults 16 to 64 years (Experimental): Adults 16 to 64 years
  Interventions: Drug: loratadine

INTERVENTIONS:
Drug: loratadine — Loratadine (SCH 29851) dry syrup 1% 5 mg/day for 4 weeks
  Other Names: Claritin; SCH 29851
  Arms: Pediatrics 3 to 6 years
Drug: loratadine — loratadine 10 mg tablet once daily for 4 weeks
  Other Names: Claritin; SCH 29851
  Arms: Pediatrics 7 to 15 years
Drug: loratadine — loratadine 10 mg tablet once daily for 4 weeks
  Other Names: Claritin; SCH 29851
  Arms: Adults 16 to 64 years

SUMMARY:
This is a post marketing study to confirm the appropriate dose of loratadine in children by obtaining drug concentration data at multiple time points per child and adult patient, after the patient receives repeated administrations of the approved dose of loratadine.

ELIGIBILITY:
Inclusion Criteria:

Patients with perennial allergic rhinitis who satisfy all of the following criteria were enrolled in the study:

* Pediatric patients between the ages of 3 and 15 years and adult patients between the ages of 16 and 64 at the time of providing informed consent.
* Outpatients of either sex.
* Pediatric patients for whom written informed consent can be obtained from the guardian before the start of the study. Adult patients from whom written informed consent can be obtained (for patients between the ages of 16 and 19, the guardian must also provide written informed consent).
* Pediatric patients who have the ability to make entries in the patient diary (Record of Drugs and Nasal Symptoms) or entry in the diary is made possible by the guardian. Adult patients who have the ability to make entries in the patient diary.
* Patients for whom treatment with loratadine monotherapy is judged appropriate based on symptoms of allergic rhinitis during the pretreatment observation period.
* Patients confirmed to be allergic to perennial allergen

Exclusion Criteria:

* Patients with a history of epileptic seizures or organic brain disorder in whom there is a possibility that epileptic seizures may be induced
* Patients with a history of hypersensitivity to any component of this drug
* Patients who are pregnant or who may be pregnant, and nursing women
* Patients with severe hepatic, renal, cardiac, or hematological disease or other serious complications and whose general condition is poor
* Patients participating in another clinical study or who have been in a clinical study within the last 30 days.
* Other patients judged inappropriate for study by the investigator or sub-investigator
* Patients allergic to pollen (cedar, mugwort, common ragweed, orchard grass, etc.) and the pollen season is during the period from 7 days before registration to the end of study drug administration
* Patients who developed diseases which might affect nasal symptoms (acute upper respiratory tract infection, acute pharyngo-laryngitis, or acute tonsillitis) in the 7 days before registration
* Patients who received treatment for allergic rhinitis in the 7 days before registration

Ages: 3 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 261 (Actual)
Dates: Start 2008-06; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Groups:
- Pediatrics 3 to 6 Years: Pediatrics 3 to 6 years of age received loratadine 5 mg/day for 28 days
- Pediatrics 7 to 15 Years: Pediatrics 7 to 15 years of age received loratadine 10 mg/day for 28 days
- Adults 16 to 64 Years: Adults 16 to 64 years of age received loratadine 10 mg/day for 28 days
Period: Overall Study
Arm/Group | Pediatrics 3 to 6 Years | Pediatrics 7 to 15 Years | Adults 16 to 64 Years
Started | 53 | 104 | 104
Completed | 53 | 104 | 103
Not Completed | 0 | 0 | 1
Not completed — Discontinued | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pediatrics 3 to 6 Years | Pediatrics 7 to 15 Years | Adults 16 to 64 Years | Total
Number analyzed (Participants) | 53 | 104 | 104 | 261
Age, Customized [Number; unit: participants]
  Between 3-6 years | 53 | 0 | 0 | 53
  Between 7 and 15 years | 0 | 104 | 0 | 104
  Between 16 - 64 years | 0 | 0 | 104 | 104
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 29 | 68 | 113
  Male | 37 | 75 | 36 | 148

OUTCOME MEASURES:

1. Primary Outcome: Mean Maximum Plasma Concentration (Cmax) of SCH 29851 (Unchanged Drug; Loratadine), SCH 34117 (Active Metabolite), and SCH 45581 (3OH-SCH 34117)
Description: SCH 29851: Two-compartment model used as basic pharmacokinetic (PK) model. Individual Cmax estimated with basic PPK parameters (apparent total body clearance (CL/F), apparent distribution volumes of central compartment (Vc/F) and peripheral compartment (Vp/F), apparent inter-compartmental clearance (Q/F), absorption rate constant (Ka), lag time, inter- and intra-individual variation) by Bayesian method. SCH 34117/SCH 45581: One-compartment model used as basic PK model. Individual Cmax was estimated with PPK parameters (above) on final model by Bayesian method.
Time Frame: After 2 and 4 weeks of treatment, and after 1 and 3 weeks of treatment if participant agreed
Population: Number of participants for SCH 29851 were 53, 104, and 104. Number of participants for SCH 34117 were 53, 102, and 104. Number of participants for SCH 44581 were 53, 99, and 104.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Pediatrics 3 to 6 Years | Pediatrics 7 to 15 Years | Adults 16 to 64 Years
Number analyzed (Participants) | 53 | 104 | 104
ng/mL
  SCH 29851 | 3.04 (1.78) | 5.54 (3.15) | 6.48 (3.28)
  SCH 34117 | 4.16 (1.26) | 4.30 (1.63) | 4.61 (1.41)
  SCH 45581 | 2.58 (0.76) | 2.56 (0.86) | 2.35 (0.54)

2. Primary Outcome: Mean Area Under the Plasma Concentration Time Curve (AUC) of SCH 29851 (Unchanged Drug), SCH 34117 (Active Metabolite), and SCH 45581 (3OH-SCH 34117)
Description: SCH 29851: Two-compartment model used as basic pharmacokinetic (PK) model. Individual AUC estimated with basic PPK parameters (apparent total body clearance (CL/F), apparent distribution volumes of central compartment (Vc/F) and peripheral compartment (Vp/F), apparent inter-compartmental clearance (Q/F), absorption rate constant (Ka), lag time, inter- and intra-individual variation) by Bayesian method. SCH 34117/SCH 45581: One-compartment model used as basic PK model. Individual AUC was estimated with PPK parameters (above) on final model by Bayesian method.
Time Frame: After 2 and 4 weeks of treatment, and after 1 and 3 weeks of treatment if participant agreed
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng•hr/mL
Arm/Group | Pediatrics 3 to 6 Years | Pediatrics 7 to 15 Years | Adults 16 to 64 Years
Number analyzed (Participants) | 53 | 104 | 104
ng•hr/mL
  SCH 29851 | 16.77 (14.87) | 26.13 (22.22) | 34.68 (37.22)
  SCH 34117 | 52.33 (15.63) | 59.52 (23.73) | 68.01 (23.33)
  SCH 45581 | 41.54 (11.43) | 42.28 (14.40) | 40.75 (9.92)

ADVERSE EVENTS:
Arm/Group | Pediatrics 3 to 6 Years | Pediatrics 7 to 15 Years | Adults 16 to 64 Years
Serious Adverse Events (participants affected / at risk) | 0/53 | 0/104 | 0/104
Other Adverse Events (participants affected / at risk) | 23/53 | 17/104 | 17/104
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Pediatrics 3 to 6 Years (N=53) | Pediatrics 7 to 15 Years (N=104) | Adults 16 to 64 Years (N=104)
Acute Tonsillitis (Infections and infestations) | 3 (3) | 0 (0) | 0 (0)
Bronchitis (Infections and infestations) | 3 (4) | 1 (1) | 0 (0)
Nasopharyngitis (Infections and infestations) | 5 (6) | 1 (1) | 9 (11)
Pharyngitis (Infections and infestations) | 9 (10) | 3 (3) | 2 (2)
White Blood Cell Count Increased (Investigations) | 3 (3) | 0 (0) | 2 (2)
Headache (Nervous system disorders) | 0 (0) | 3 (3) | 6 (7)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 5 (13) | 9 (11) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The investigator (sub-investigator) will disclose the results and knowledge obtained through this study after discussion with the Sponsor and approval is obtained from the Sponsor.

If the investigator (sub-investigator) is to present the results obtained from this study at a medical conference or medical journal, approval of the Sponsor must be obtained beforehand